CLINICAL TRIAL: NCT05057429
Title: A Bioelectric Dressing for Post De-Roofing Treatment of Hidradenitis Suppurativa (HS)
Brief Title: A Bioelectric Dressing for Post De-Roofing Treatment of HS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Vomaris Innovations (Industry)
Responsible Party: Principal Investigator, Hadar Lev-Tov, Assistant Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210621
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-07

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bioelectric Dressing on the Right Armpit and Standard Gauze Dressing on the Left Armpit (Experimental): Participants undergoing standard of care deroofing surgery will be randomized to receive the bioelectric dressing for up to 8 weeks on the right armpit and will receive the standard gauze dressing for up to 8 weeks on the left armpit.
  Interventions: Device: Procellera Bioelectric Dressing; Other: Standard Gauze Dressing
- Bioelectric Dressing on the Left Armpit and Standard Gauze Dressing on the Right Armpit (Experimental): Participants undergoing standard of care deroofing surgery will be randomized to receive the bioelectric dressing for up to 8 weeks on the left armpit and will receive the standard gauze dressing for up to 8 weeks on the right armpit.
  Interventions: Device: Procellera Bioelectric Dressing; Other: Standard Gauze Dressing

INTERVENTIONS:
Device: Procellera Bioelectric Dressing — Procellera is single layer, broad-spectrum antimicrobial wound dressing. Embedded in the dressing are microcell batteries made of elemental silver and zinc applied in a dot-matrix pattern. The bioelectric dressing will be applied to surgical site wound with a hydrogel.
Other: Standard Gauze Dressing — Standard of care non-adherent gauze dressing will be applied to surgical site with vaseline.

SUMMARY:
The primary purpose of this study is to test if the use of a bioelectric dressing can improve healing after a surgical procedure called de-roofing.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old and older.
* Have diagnosis of HS confirmed by a dermatologist
* Have at least two ancillary tunnels in separate anatomical sites
* Able to provide informed consent

Exclusion Criteria:

* Individuals who are not yet adults
* Subject is allergic to any of the materials and dressings involved in the procedures
* Women known to be pregnant
* Prisoners
* Subjects, who in the opinion of the PI, cannot comply with hope application of the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Healing Rate | Up to 8 weeks
  The healing rate of post-surgical wounds will be reported as the area reduction in cm^2/per day.

SECONDARY OUTCOMES:
Average time to complete healing | Up to 8 weeks
  The average time, measured in days, to complete healing as assessed by treating physician will be reported
Number of subjects with complete healing | Up to 8 weeks
  The number of subjects with complete post-surgical site healing, as evaluated by treating physician, will be reported.
Number of subjects with nodule and/or tunnel recurrence | Up to 8 weeks
  The number of subjects with nodule and/or tunnel recurrence, as evaluated by treating physician, will be reported.
Average pain as assessed by the Numerical Rating Scale (NRS) | Up to 8 weeks
  The average pain will be measured using the NRS with scores ranging from 0-10 with the higher score indicating more severe pain.
Number of subjects with tenderness at surgical sites | Up to 8 weeks
  The number of subjects with tenderness at surgical sites, as evaluated by treating physician, will be reported.
Quality of post-surgical scars as measured by the Hurley Stage score | Up to 8 weeks
  The Hurley score is staged as: 1 (single or multiple abscesses without sinus tract formation or scarring); 2 (recurrent abscesses with one or more sinus tracts and scarring widely separated by normal skin); 3 (diffuse involvement with multiple sinus tracts and no intervening normal skin)
Amount of exudate at surgical site | Up to 8 weeks
  The amount of exudate at surgical site will be evaluated using a 5 point Likert scale from 0 (Dry) to 4 (Leaking).
Shoulder range of motion | Up to 8 weeks
  Shoulder range of motion will be measured using a goniometer
Number of dressings used through to healing day | Up to 8 weeks
  The number of dressings used through to healing day will be reported
Pain after procedure as assessed by the NRS | Day 2 (24 hours post procedure)
  The average pain will be measured using the NRS with scores ranging from 0-10 with the higher score indicating more severe pain.
Days of work lost | Up to 8 weeks
  Participants reported days of work lost due to the procedure will be reported
Change in Quality of Life as measured by the DLQI | Baseline, Up to 8 weeks
  Dermatology Life Quality Index (DLQI) has a total score ranging from 0 to 30 with the lower score indicating higher health related quality of life
Tissue analysis of microbiome | Up to 8 weeks
  As measured by quantitative 16s rDNA Polymerase Chain Reaction for bacterial enumeration from punch biopsy and biofilm samples.

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Lev-Tov, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No